CLINICAL TRIAL: NCT01875003
Title: A Study of Lebrikizumab in Adolescent Participants With Uncontrolled Asthma Who Are on Inhaled Corticosteroids and a Second Controller Medication
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WB28183; 2012-000180-25 (EudraCT Number)
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — lebrikizumab; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes

ARMS (3):
- Lebrikizumab High (Experimental): Participants with uncontrolled asthma on ICS therapy (total daily dose of 500-2000 micrograms [mcg] of fluticasone propionate dry powder inhaler [DPI] or equivalent) and a second controller medication, will receive SC injection of lebrikizumab (high dose) Q4W for 52 weeks during placebo-controlled period and up to 76 weeks or 104 weeks for participants who will be willing to take part in optional active-treatment extension period.
  Interventions: Drug: Lebrikizumab; Drug: Standard of Care
- Lebrikizumab Low (Experimental): Participants with uncontrolled asthma on ICS therapy (total daily dose of 500-2000 mcg of fluticasone propionate DPI or equivalent) and a second controller medication, will receive SC injection of lebrikizumab (low dose) Q4W for 52 weeks during placebo-controlled period and up to 76 weeks or 104 weeks for participants who will be willing to take part in optional active-treatment extension period.
  Interventions: Drug: Lebrikizumab; Drug: Standard of Care
- Placebo (Placebo Comparator): Participants with uncontrolled asthma on ICS therapy (total daily dose of 500-2000 mcg of fluticasone propionate DPI or equivalent) and a second controller medication, will receive SC injection of lebrikizumab matching placebo Q4W for 52 weeks during placebo-controlled period and then SC injection of lebrikizumab at high or low dose will be administered from Weeks 52 to 76 or 104 to participants who are willing to take part in optional active-treatment extension period.
  Interventions: Drug: Lebrikizumab; Drug: Placebo; Drug: Standard of Care

INTERVENTIONS:
Drug: Lebrikizumab — Lebrikizumab will be administered as SC injection at high or low dose Q4W.
Drug: Placebo — Lebrikizumab matching placebo will be administered as SC injection Q4W.
  Arms: Placebo
Drug: Standard of Care — Participants will continue to receive ICS therapy (total daily dose of 500-2000 mcg fluticasone propionate DPI or equivalent) along with at least one second controller medications (e.g. long-acting beta agonists [LABAs], leukotriene receptor antagonists (LTRAs), long-acting muscarinic antagonists (LAMAs), or theophylline) as standard of care.

SUMMARY:
This randomized, multicenter, double-blind, placebo-controlled, parallel-group study will evaluate the efficacy, safety, and tolerability of lebrikizumab in adolescent participants with asthma whose disease remains uncontrolled despite daily treatment with inhaled corticosteroids (ICS) therapy and at least one second controller medication. Participants will be randomized in a 1:1:1 ratio to receive double-blind treatment with either lebrikizumab ('High' or 'Low') or placebo, administered as subcutaneous (SC) every 4 weeks (Q4W) for 52 weeks, in addition to their standard-of-care therapy. This will be followed by an optional 52-week double-blind active-treatment extension. The anticipated time on study treatment is up to 104 weeks. Participants who complete the study to Week 104, discontinue prematurely or decide not to take part in the optional active-treatment extension will transition to the 20-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosis for greater than or equal to (>/=) 12 months prior to Visit 1
* Bronchodilator response during screening
* Pre-bronchodilator FEV1 of 40 percent (%) - 90% predicted at both Visits 2 and 3
* On high dose ICS therapy for >/= 6 months prior to Visit 1
* On an eligible second controller medication for 6 months prior to Visit 1
* Uncontrolled asthma as defined by the protocol both during screening and at the time of randomization
* Demonstrated adherence with controller medication during the screening period

Exclusion Criteria:

* History of severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the lebrikizumab injection
* Maintenance oral corticosteroid therapy within 3 months prior to Visit 1
* Treatment with systemic (oral, intravenous [IV], or intramuscular [IM]) corticosteroids within 4 weeks prior to Visit 1 or during the screening period
* Treatment with intra-articular corticosteroids within 4 weeks prior to Visit 1 or during the screening period or anticipated need for intra-articular corticosteroids during the course of the study
* Infection that meets the following criteria: Any infection requiring hospital admission or requiring treatment with IV or IM antibiotics within 4 weeks prior to Visit 1 or during screening; any active infection that required treatment with oral antibiotics within 2 weeks prior to Visit 1 or during screening; upper or lower respiratory tract infection within 4 weeks prior to Visit 1 or during screening; active parasitic infection or Listeria monocytogenes infection within 6 months prior to Visit 1 or during screening
* History of active tuberculosis requiring treatment
* Known immunodeficiency, including, but not limited to, human immunodeficiency virus (HIV) infection
* Evidence of acute or chronic hepatitis or known liver cirrhosis
* History of cystic fibrosis, bronchiectasis, and/or other clinically significant lung disease other than asthma
* Diagnosis or history of malignancy or current evaluation for potential malignancy
* Current smoker or former smoker with a history of greater than (>) 10 pack-years
* History of alcohol or drug abuse
* Past and/or current use of any anti- interleukin (IL) -13 or anti-IL-4/IL-13 therapy, including lebrikizumab
* Use of other monoclonal antibody therapy, including omalizumab, within 6 months or 5 drug half-lives (whichever is longer) prior to Visit 1
* Initiation of or change in allergen immunotherapy within 3 months prior to Visit 1 or during screening
* History of bronchial thermoplasty

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 348 (Actual)
Dates: Start 2013-08-31 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
Rate of Asthma Exacerbations During the 52-Week Placebo-Controlled Period | Baseline up to Week 52
Percentage of Participants With Adverse Events (AEs) or Serious AEs | Baseline up to Week 124
Percentage of Participants With Anti-Therapeutic Antibodies to Lebrikizumab | Baseline up to Week 124 (assessed at Baseline, Weeks 4, 12, 24, 36, 52, 76, 104, 112, and 124 or at early termination [up to 108 weeks])

SECONDARY OUTCOMES:
Change from Baseline in Pre-Bronchodilator Forced Expiratory Volume in 1 second (FEV1) at Week 52 | Baseline , Week 52
Time to First Asthma Exacerbation | Baseline up to 52 weeks
Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO) at Week 52 | Baseline , Week 52
Change From Baseline in Standardized Asthma Quality of Life Questionnaire for 12 years and Older (AQLQ + 12) at Week 52 | Baseline, Week 52
Change From Baseline in Asthma Rescue Medication Use at Week 52 | Baseline, Week 52
Rate of Urgent Asthma-Related Health Care Utilization | Baseline up to 52 weeks
Injection Acceptability Questionnaire (IAQ) Score | Baseline up to Week 104

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (165):
- United States (43):
  - Allergy Associates of Tucson, Tucson, Arizona
  - Kaiser Permanente Los Angeles, Los Angeles, California
  - Southern California Research Center, Mission Viejo, California
  - Allergy & Asthma Consultants, Redwood City, California
  - Dignity Health Medical Foundation, Sacramento, California
  - Bensch Research Associates, Stockton, California
  - Allergy & Asthma Medical Group; Clinical Research Division, Walnut Creek, California
  - Colorado Children's Hospital; The Breathing Institute, Aurora, Colorado
  - IMMUNOe International Research Centers, Centennial, Colorado
  - Asthma & Allergy; Associates, P.C., Colorado Springs, Colorado
  - National Jewish Medical and Research Center, Denver, Colorado
  - Abel and Buchheim, Miami, Florida
  - Compass Research East, LLC, Orlando, Florida
  - Sarasota Clinical Research, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Brookstone Clinical Res Ctr, Columbus, Georgia
  - Georgia Pain Clinic, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - The Clinical Research Center, Shiloh, Illinois
  - Riley Hospital for Children; Pediatric Nephrology, Indianapolis, Indiana
  - Abraham Research PLLC, Florence, Kentucky
  - Breathe America Shreveport Inc, Shreveport, Louisiana
  - Asthma, Allergy & Sinus Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Univ of Michigan Medical Ctr, Ann Arbor, Michigan
  - Cardinal Glennon Child's Hosp; Endrocrinology, St Louis, Missouri
  - Parikh Institute for Research LLC, New Jersey, New Jersey
  - University of New Mexico; School of Med, Albuquerque, New Mexico
  - Parikh Institute for Research LLC, New York, New York
  - Urban Health Plan, Inc., The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Promedica Toledo Children's Hospital, Toledo, Ohio
  - Bend Memorial Clinic, Bend, Oregon
  - Allergy, Asthma, & Dermatology Research Center, Llc, Lake Oswego, Oregon
  - Clinical Research Inst. of Southern Oregon, Pc, Medford, Oregon
  - TTS Research, Boerne, Texas
  - Allergy & Asthma Research Center of El Paso, El Paso, Texas
  - Allergy & Asthma Res Ctr PA, San Antonio, Texas
  - South Texas Allergy and Asthma Medical Professionals, San Antonio, Texas
  - Bridgerland Clinical Research, North Logan, Utah
  - O & O Alpan, LLC, Fairfax, Virginia
  - Bellingham Asthma, Allergy & Immunology, Bellingham, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (12):
  - Centro Médico Vitae, Buenos Aires
  - Fundación Faicep, Buenos Aires
  - Fundacion Cidea, Buenos Aires
  - INAER, Buenos Aires
  - Instituto Respirar, Mendoza
  - INSARES, Mendoza, Mendoza City
  - Centro Respiratorio Infantil, Rosario
  - Investigaciones en Patologias Respiratorias, San Miguel de Tucumán
  - Centro Integral de Medicina Respiratoria (CIMER), San Miguel de Tucumán
  - Instituto Del Buen Aire, Santa Fe
  - Sanatorio Británico de Rosario, Santa Fé
  - CEMER Centro Médico de Enfermedades Respiratorias, Vicente López
- Brazil (8):
  - Centro de Referencia em Enfermidades Respiratorias e Alergia - CEAR, Salvador, Estado de Bahia
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina do ABC - FMABC, Santo André, São Paulo
  - Pesquisare Saúde Sociedade Simples, Santo André, São Paulo
  - Hospital Alemao Oswaldo Cruz; Pesquisa Clinica, São Paulo, São Paulo
  - Instituto de Pesquisa Clínica e Medicina Avançada Ltda, São Paulo, São Paulo
  - CMPC/Clinica de Alergia Martti Antila, Sorocaba, São Paulo
- Canada (3):
  - Dr. Tharwat A. Fera Inc., Vancouver, British Columbia
  - Brian Lyttle's Private Practice, London, Ontario
  - Centre de Recherche Applique En Allergie de Quebec, Québec, Quebec
- Colombia (2):
  - Hospital Santa Clara, Bogotá
  - Hospital Pablo Tobon Uribe, Medellin-Antioquia
- Czechia (2):
  - Hofstetr Alois MUDr. s.r.o., Jihlava
  - Alergologie Teplice, s.r.o., Teplice
- France (4):
  - Groupe Hospitalier Pellegrin; Pharmacie, Bordeaux
  - Groupe Hospitalier Necker Enfants Malades, Paris
  - Hopital Armand Trousseau, Paris
  - Hopital Charles Nicolle; cic, Rouen
- Germany (3):
  - Universitaetsklinikum Frankfurt, Frankfurt
  - Evangelisches Krankenhaus Hamm, Hamm
  - Praxis Dr. med. Jan Feimer, München
- Hungary (7):
  - Semmelweis Egyetem, Budapest
  - Heim Pál Gyermekkórház, Budapest
  - Kenezy Korhaz Rendelointezet, Debrecen
  - Borsod-Abaúj-Zemplén Megyei Kórház és Egyetemi Oktató Kórház, Miskolc
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
  - Papp és Társa Bt., Szigetvár
  - Tudogyogyintezet Torokbalint, Törökbálint
- Israel (5):
  - Barzilai Medical Center, Ashkelon
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (4):
  - Azienda Policlinico Umberto I; Dipartimento Integrato di Pediatria e Neuropsichiatria Infantile, Rome, Lazio
  - Ospedale Pediatrico Bambino Gesu, Rome, Lazio
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy
  - Azienda Ospedaliero - Universitaria Policlinico - Vittorio Emanuele, Catania, Sicily
- Japan (2):
  - National Hospital Organization Mie Hospital, Tsu
  - National Hospital Organization Shimoshizu National Hospital, Yotsukaidō
- Mexico (8):
  - Grupo Medico Camino, DF
  - Instituto Jalisciense de Investigacion Clinica S.A. de C.V., Guadalajara
  - Centro de Investigacion Medico Biologico y Terapia Avanzada, S.C., Guadalajara
  - Unidad Medica de Occidente, Guadalajara
  - Instituto Nacional de Pediatría, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio González; Enfermedades Pulmonares Crónicas, Monterrey
  - Unidad de Investigacion Clinica En Medicina (Udicem) S.C., Monterrey
  - Consultorio Especialidad Alergologia Pediatrica, Villahermosa
- Peru (6):
  - Hospital Dos de Mayo; Parque Historia De la Medicina Peruana S/n, Lima
  - Hospital Nacional Luis N Saenz PNP, Lima
  - Clinica Internacional, Lima
  - Centro de Investigación Ricardo Palma, Lima
  - Clinica Anglo Americana, Lima
  - Clinica San Borja, Lima
- Poland (8):
  - Prywatna Praktyka Lekarska, Bialystok
  - Malopolskie Centrum Alergologii, Krakow
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika w Lodzi, Lodz
  - Centrum Alergologii NZOZ, Lublin
  - Centrum Alergologii Teresa Hofman, Poznan
  - ALERGO-MED Specjalistyczna Przychodnia Lekarska Sp. z o. o, Tarnów
  - Klinika Chorób Wewnetrznych i Alergologii MSW, Warsaw
- Portugal (4):
  - Hospital Infante D. Pedro; Servico de Imunoalergologia, Aveiro
  - Hospital Particular do Algarve - Unidade de Faro, Faro
  - Hospital Dona Estefania; Servico de Imunoalergologia, Lisbon
  - Hospital CUF Porto; Servico de Imunoalergologia, Senhora Da Hora - Porto
- Slovakia (3):
  - Alersa, Košice
  - ALERGOMEA s.r.o., Lučenec
  - Imunoalergologia Dzurilla s.r.o., Nitra
- South Africa (9):
  - Uni of Cape Town Lung Inst., Cape Town
  - Westville Hospital, Durban
  - Sebastian Peter, Durban
  - WWCT Lakeview Hospital, Johannesburg
  - Medicross Sophiatown, Johannesburg
  - GCT Mercantile; Clinical Research Centre, Port Elizabeth
  - Bothe ke Bontle Health Services, Pretoria
  - Soweto Clinical Trial Centre, Soweto
  - Limpopo Clinical Research Initiative; Tamboti Medical Centre, Tabazimbi
- South Korea (3):
  - Inha University Hospital, Incheon
  - Severance Hospital, Yonsei University Health System, Seoul
  - KyungHee Medical Center, Seoul
- Spain (9):
  - Hospital Universitario Germans Trias i Pujol; Servicio de Farmacia, Badalona, Barcelona
  - Hospital Sant Joan De Deu, Esplugues de Llobregas, Barcelona
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital de Manises, Manises, Valencia
  - Hospital Quiron Teknon, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Clínica Dr. Lobatón, Cadiz
  - Clinica Ojeda de Asma Y Alergia, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
- Taiwan (5):
  - Chung Shan M. U. H., Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung Univ Hosp, Tainan
  - Chang Gung Memorial Hospital, Taoyuan District
- Ukraine (7):
  - Municipal Medical Institution; Chernivtsi Regional Children's Hospital, Chernivtsi
  - Public Institution City Clinical Hospital # 6 of Dnipropetrovsk Regional Board, Dnipro
  - State Institution of Pediatrics Obstetrics and Gynecology of NAMSU, Kiev
  - Municipal Institution "Kryvyi Rih City Clinical Hospital #8" of Dnipropetrovsk Regional Council, Kryvyi Rih
  - SI National Institute of Phthisiology and Pulmonology n.a. F.G.Yanovskyi under NAMS of Ukraine, Kyiv
  - SI Research Centre of Radiation Medicine of AMSU, Kyiv
  - Municipal Institution Zaporizhzhya Regional Clinical Child Hospital, Zaporizhzhya
- United Kingdom (8):
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - Birmingham Heartlands Hospital, Birmingham
  - Dumfries and Galloway Royal Infirmary; Department of Paediatrics, Dumfries
  - Royal Hospital For Children, Glasgow
  - University of Leicester, Leicester
  - Royal Brompton Hospital; Respiratory Department, London
  - Sheffield Childrens Hospital, Sheffield
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Szefler SJ, Roberts G, Rubin AS, Zielen S, Kuna P, Alpan O, Anzures-Cabrera J, Chen Q, Holweg CTJ, Kaminski J, Putnam WS, Matthews JG, Kamath N. Efficacy, safety, and tolerability of lebrikizumab in adolescent patients with uncontrolled asthma (ACOUSTICS). Clin Transl Allergy. 2022 Jul 14;12(7):e12176. doi: 10.1002/clt2.12176. eCollection 2022 Jul. PMID 35846226